CLINICAL TRIAL: NCT00150709
Title: A Multi-Center, Open-Label, Long-Term, Follow-Up Study Of The Safety And Efficacy Of Levetiracetam (Ucb L059) In Children With Epilepsy
Brief Title: A Study Of The Safety And Efficacy Of Levetiracetam (Keppra®) (Ucb L059) In Children With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N157
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-06

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Pediatric; Partial onset epilepsy; Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- N159 PBO/LEV (Experimental): Subjects had previously participated in study N159 in which they had received Placebo (PBO).
  Interventions: Drug: Levetiracetam
- N159 LEV/LEV (Experimental): Subjects had previously participated in study N159 in which they had received Levetiracetam (LEV).
  Interventions: Drug: Levetiracetam
- N01010+N151 LEV/LEV (Experimental): Subjects had previously participated in study N01010 or study N151 in which they had received Levetiracetam (LEV).
  Interventions: Drug: Levetiracetam
- N01052 LEV/LEV (Experimental): Subjects had previously participated in study N01052 in which they had received Levetiracetam (LEV).
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — * Pharmaceutical form: Oral tablets and oral solution
  * Route of administration: Oral use
  Other Names: Keppra

SUMMARY:
Open-label study to allow pediatric patients who have participated in prior Levetiracetam (Keppra®) studies to continue their treatment with adequate monitoring and standardized follow-up care until Levetiracetam (Keppra®) is approved for use in children or until the completion of the development program for pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Have completed Study N151, or any other applicable pediatric trials of Levetiracetam (Keppra®)
* Be a patient for whom the treatment of Levetiracetam (Keppra®) would be of potential benefit such that the patient/parent(s)/legal guardian and the Investigator agree to continue treatment.

Exclusion Criteria:

* Not be on a ketogenic diet (during the course of this study).
* Not have seizures too close together to accurately count (i.e., the patient's seizures must be countable).

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 1998-01-26 (Actual); Primary Completion 2006-01-25 (Actual); Study Completion 2006-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 1998 and concluded in January 2006.
Pre-assignment Details: Participant Flow refers to the Intention-to-treat (ITT) Set.
Period: Overall Study
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Started | 79 | 89 | 41 | 14
Completed | 24 | 27 | 17 | 6
Not Completed | 55 | 62 | 24 | 8
Not completed — Protocol Violation | 7 | 8 | 3 | 1
Not completed — Adverse Event | 8 | 2 | 2 | 3
Not completed — Lack of Efficacy | 6 | 11 | 9 | 0
Not completed — Withdrawal by Subject | 7 | 10 | 5 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 1
Not completed — Site/Investigator discontinued the study | 5 | 5 | 2 | 0
Not completed — Decision of parent(s) | 1 | 2 | 0 | 0
Not completed — Decision of parent(s) and investigator | 3 | 0 | 0 | 0
Not completed — Loss/ incompleteness of efficacy | 12 | 12 | 2 | 2
Not completed — Investigator decision | 1 | 0 | 0 | 1
Not completed — Subject relocated | 2 | 2 | 1 | 0
Not completed — Subject continues Keppra through prescriptions | 0 | 4 | 0 | 0
Not completed — Convenience | 0 | 1 | 0 | 0
Not completed — Subject entered new drug study | 0 | 1 | 0 | 0
Not completed — Subject to undergo surgery for seizures | 0 | 1 | 0 | 0
Not completed — Lack of ease of swallowing | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Intention-to-treat (ITT) Set which consisted of all subjects who took at least one dose of levetiracetam in study N157 excluding subjects from one site due to the unreliability of the data reported.
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV | Total Title
Number analyzed (Participants) | 79 | 89 | 41 | 14 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 79 | 89 | 41 | 14 | 223
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.88 (3.46) | 10.61 (3.24) | 10.07 (2.20) | 1.62 (1.16) | 9.68 (3.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 16 | 7 | 105
  Male | 36 | 50 | 25 | 7 | 118

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Partial Onset (Type I) Seizure Frequency Per Week Over Time During the Treatment Period
Description: Percentage change from Baseline of partial onset (Type I) seizure frequency over the Treatment Period standardized to 1 week Period. According to the ILAE 1981 classification, seizures can be classified into one of the following three groups: Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures). Negative values indicate an improvement from Baseline.
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: Only subjects with valid data for Partial (Type I) seizure frequency at both baseline and during the treatment period are included in the analysis. The data for N01052 LEV/LEV arm was not available as the prior study N01052 did not collect baseline seizure information and therefore N01052 study participants were excluded systematically due to missing baseline measurements.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 87 | 41 | 0
percentage of change | -66.4 [-90.0 to -22.3] | -47.8 [-76.2 to -25.4] | -66.4 [-93.6 to -5.6] |

2. Primary Outcome: Percentage Change From Baseline in Total (Type I, II, III) Seizure Frequency Per Week Over Time During the Treatment Period
Description: Percentage change from Baseline in total (type I, II, III) seizure frequency over the Treatment Period standardized to 1 week Period. Seizures were categorized in Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures) according to the ILAE 1981 classification. Negative values indicate an improvement from Baseline.
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: Only subjects with valid data for total (Type I, II, III) seizure frequency at both baseline and during the treatment period are included in the analysis. The data for N01052 LEV/LEV arm was not available as the prior study N01052 did not collect baseline seizure information and therefore N01052 study participants were excluded systematically due to missing baseline measurements.
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 88 | 41 | 0
percentage of change | -66.4 [-90.0 to -25.2] | -45.7 [-73.6 to -17.4] | -65.9 [-93.1 to -5.6] |

3. Secondary Outcome: Absolute Change From Baseline in Partial Onset (Type I) Seizure Frequency Over Time During the Treatment Period
Description: Absolute change from Baseline of Partial onset (Type I) seizure frequency over the Treatment Period standardized to 1 week Period. According to the ILAE 1981 classification, seizures can be classified into one of the following three groups: Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures). Negative values indicate an improvement from Baseline.
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: Only subjects with valid data for Partial Onset (Type I) seizure frequency at both baseline and during the treatment period are included in the analysis. The data for N01052 LEV/LEV arm was not available as the prior study N01052 did not collect baseline seizure information and therefore N01052 study participants were excluded systematically due to missing baseline measurements.
Measure: Median (Inter-Quartile Range); unit: partial seizure frequency per week
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 87 | 41 | 0
partial seizure frequency per week | -2.1 [-7.4 to -0.3] | -1.6 [-6.6 to -0.6] | -1.5 [-7.4 to 0.0] |

4. Secondary Outcome: Absolute Change From Baseline in Total (Type I, II, III) Seizure Frequency Per Week Over Time During the Treatment Period
Description: Absolute change from Baseline in total (type I, II, III) seizure frequency over the Treatment Period standardized to 1 week period. Seizures were categorized in Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures) according to the ILAE 1981 classification. Negative values indicate improvement from Baseline.
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: partial seizure frequency per week
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 88 | 41 | 0
partial seizure frequency per week | -2.1 [-7.4 to -0.6] | -1.5 [-6.4 to -0.5] | -1.1 [-7.3 to 0.0] |

5. Secondary Outcome: At Least 50% Responder Rate in Partial Onset (Type I) Seizure Frequency From Baseline Per Week During the Treatment Period
Description: At least 50% responder rate in Partial Onset (Type I) Seizure Frequency per Week over the Treatment Period is defined as the percentage of subjects with a reduction from baseline in Partial Onset (Type I) seizure frequency of at least 50%. According to the ILAE 1981 classification, seizures can be classified into one of the following three groups: Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures).
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: Only subjects who have a baseline greater than zero for partial onset (Type I) seizures and valid N157 seizure information are included in the analysis. The data for N01052 LEV/LEV arm was not available as the prior study N01052 did not collect baseline seizure information and therefore N01052 study participants were excluded systematically due to missing baseline measurements.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 77 | 86 | 37 | 0
percentage of participants | 58.4 | 47.7 | 62.2 |

6. Secondary Outcome: At Least 50% Responder Rate in Total (Type I, II, III) Seizure Frequency From Baseline Per Week During the Treatment Period
Description: At least 50% responder rate in total (Type I, II, III) Seizure Frequency per Week over the Treatment Period is defined as the percentage of subjects with a reduction from baseline in total (Type I, II, III) seizure frequency of at least 50%. Seizures were categorized in Type I (partial onset seizures), Type II (generalized seizures) and Type III (unclassified seizures) according to the ILAE 1981 classification.
Time Frame: During the Treatment Period (an average of 2 years), compared to Baseline
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 77 | 88 | 37 | 0
percentage of participants | 58.4 | 46.6 | 62.2 |

7. Secondary Outcome: Number of Subjects Who Are Seizure-free for at Least 7 Days During the Treatment Period
Description: A day was considered seizure-free if no seizures were reported for 24 hours.
Time Frame: During the Treatment Period (an average of 2 years)
Measure: Count of Participants; unit: Participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
Participants | 74 | 73 | 40 | 10

8. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (Day 0)
Description: A time interval was considered seizure-free if no seizures were reported in that time interval. The Treatment Period consisted of a 6-week Titration Phase and a Maintenance Phase lasting until market approval or completion of development of levetiracetam for the pediatric indication.
Time Frame: Day 0 (beginning day of the maintenance phase)
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 74.0 | 64.0 | 75.0 | 38.5

9. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (Day 1 - <= 2 Months)
Description: as for outcome 8
Time Frame: Day 1 - <= 2 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 16.4 | 15.1 | 27.5 | 23.1

10. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 2 Months - <= 4 Months)
Description: as for outcome 8
Time Frame: > 2 months - <= 4 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 12.3 | 12.8 | 17.5 | 23.1

11. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 4 Months - <= 6 Months)
Description: as for outcome 8
Time Frame: > 4 months - <= 6 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 11.0 | 9.3 | 15.0 | 11.5

12. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 6 Months - <= 8 Months)
Description: as for outcome 8
Time Frame: > 6 months - <= 8 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 8.2 | 4.7 | 12.5 | 11.5

13. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 8 Months - <= 10 Months)
Description: as for outcome 8
Time Frame: > 8 months - <= 10 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 5.5 | 3.5 | 10.0 | 11.5

14. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 10 Months - <= 12 Months)
Description: as for outcome 8
Time Frame: > 10 months - <= 12 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 1.4 | 3.5 | 7.5 | 11.5

15. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 12 Months - <= 14 Months)
Description: as for outcome 8
Time Frame: > 12 months - <= 14 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 1.4 | 2.3 | 5.0 | 11.5

16. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 14 Months - <= 16 Months)
Description: as for outcome 8
Time Frame: > 14 months - <= 16 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 1.4 | 2.3 | 5.0 | 11.5

17. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 16 Months - <= 18 Months)
Description: as for outcome 8
Time Frame: > 16 months - <= 18 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 1.4 | 2.3 | 2.5 | 11.5

18. Secondary Outcome: Cumulative Percentage of Subjects Who Are Continuously Seizure Free by Time Interval (> 18 Months - <= 20 Months)
Description: as for outcome 8
Time Frame: > 18 months - <= 20 months of the Maintenance Phase
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
percentage of participants | 1.4 | 2.3 | 2.5 | 11.5

19. Secondary Outcome: Number of Seizures by Type During the Treatment Period
Description: Number of following seizure types were assessed: Total seizures (Type I, II, III), Total Type I seizures, Total Type II seizures, Total Type III seizures
Time Frame: During the Treatment Period (an average of 2 years)
Measure: Number; unit: seizures
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 79 | 89 | 41 | 14
seizures
  Total seizures (Type I, II, III) | 42132 | 70121 | 24232 | 19914
  Total Type I seizures | 39147 | 57464 | 24089 | 13675
  Total Type II seizures | 2142 | 12656 | 142 | 6239
  Total Type III seizures | 843 | 1 | 1 | 0

20. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 1
Description: Disease evolution compared to the last visit was evaluated by the investigator applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening, not done. The Global Evaluation Scale (GES) is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit). The reference time point for Visit 1 is in the respective feeder study of the participant.
Time Frame: Visit 1 (Screening Visit (Week 0))
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 89 | 41 | 14
percentage of participants
  Marked improvement | 7.7 | 11.2 | 29.3 | 0.0
  Moderate improvement | 21.8 | 18.0 | 12.2 | 0.0
  Slight improvement | 12.8 | 24.7 | 19.5 | 0.0
  No change | 47.4 | 40.4 | 26.8 | 100.0
  Slight worsening | 5.1 | 5.6 | 12.2 | 0.0
  Moderate worsening | 3.8 | 0.0 | 0.0 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 1.3 | 0.0 | 0.0 | 0.0

21. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 1
Description: Disease evolution compared to the last visit was evaluated by the investigator applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening, not done. The Global Evaluation Scale (GES) is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit).
Time Frame: Titration Visit 1 (Week 2)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis. The data for 'N01010+N151 LEV/LEV' and 'N01052 LEV/LEV' arms was not available as the Titration Visit 1 was required only for subjects previously enrolled in N159.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 74 | 82 | 0 | 0
percentage of participants
  Marked improvement | 14.9 | 6.1 |  |
  Moderate improvement | 14.9 | 14.6 |  |
  Slight improvement | 32.4 | 18.3 |  |
  No change | 33.8 | 47.6 |  |
  Slight worsening | 4.1 | 9.8 |  |
  Moderate worsening | 0.0 | 2.4 |  |
  Marked worsening | 0.0 | 0.0 |  |
  Not done | 0.0 | 1.2 |  |

22. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 2
Description: Disease evolution compared to the last visit was evaluated by the investigator applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening, not done. The GES is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit).
Time Frame: Titration Visit 2 (Week 4)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis. The data for 'N01010+N151 LEV/LEV' and 'N01052 LEV/LEV' arms was not available as the Titration Visit 2 was required only for subjects previously enrolled in N159.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 75 | 84 | 0 | 0
percentage of participants
  Marked improvement | 10.7 | 13.1 |  |
  Moderate improvement | 20.0 | 8.3 |  |
  Slight improvement | 20.0 | 15.5 |  |
  No change | 37.3 | 46.4 |  |
  Slight worsening | 9.3 | 11.9 |  |
  Moderate worsening | 2.7 | 2.4 |  |
  Marked worsening | 0.0 | 0.0 |  |
  Not done | 0.0 | 2.4 |  |

23. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 3
Description: as for outcome 22
Time Frame: Titration Visit 3 (Week 6)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis. The data for 'N01010+N151 LEV/LEV' and 'N01052 LEV/LEV' arms was not available as the Titration Visit 3 was required only for subjects previously enrolled in N159.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 67 | 73 | 0 | 0
percentage of participants
  Marked improvement | 10.4 | 4.1 |  |
  Moderate improvement | 14.9 | 8.2 |  |
  Slight improvement | 17.9 | 21.9 |  |
  No change | 41.8 | 47.9 |  |
  Slight worsening | 7.5 | 9.6 |  |
  Moderate worsening | 4.5 | 4.1 |  |
  Marked worsening | 0.0 | 1.4 |  |
  Not done | 3.0 | 2.7 |  |

24. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 2
Description: as for outcome 22
Time Frame: Visit 2 (Month 2)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 73 | 84 | 39 | 12
percentage of participants
  Marked improvement | 4.1 | 8.3 | 20.5 | 16.7
  Moderate improvement | 15.1 | 14.3 | 20.5 | 16.7
  Slight improvement | 26.0 | 17.9 | 25.6 | 25.0
  No change | 34.2 | 46.4 | 28.2 | 16.7
  Slight worsening | 15.1 | 8.3 | 2.6 | 0.0
  Moderate worsening | 2.7 | 2.4 | 2.6 | 8.3
  Marked worsening | 1.4 | 2.4 | 0.0 | 16.7
  Not done | 1.4 | 0.0 | 0.0 | 0.0

25. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 3
Description: as for outcome 22
Time Frame: Visit 3 (Month 4)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 68 | 77 | 38 | 10
percentage of participants
  Marked improvement | 4.4 | 6.5 | 15.8 | 20.0
  Moderate improvement | 7.4 | 3.9 | 15.8 | 0.0
  Slight improvement | 20.6 | 14.3 | 26.3 | 30.0
  No change | 41.2 | 50.6 | 34.2 | 40.0
  Slight worsening | 20.6 | 20.8 | 7.9 | 10.0
  Moderate worsening | 5.9 | 3.9 | 0.0 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

26. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 4
Description: as for outcome 22
Time Frame: Visit 4 (Month 6)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 63 | 75 | 35 | 10
percentage of participants
  Marked improvement | 4.8 | 4.0 | 14.3 | 10.0
  Moderate improvement | 6.3 | 10.7 | 17.1 | 10.0
  Slight improvement | 23.8 | 28.0 | 8.6 | 10.0
  No change | 42.9 | 34.7 | 42.9 | 60.0
  Slight worsening | 12.7 | 17.3 | 14.3 | 10.0
  Moderate worsening | 7.9 | 4.0 | 2.9 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 1.6 | 1.3 | 0.0 | 0.0

27. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 5
Description: as for outcome 22
Time Frame: Visit 5 (Month 9)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 59 | 65 | 32 | 9
percentage of participants
  Marked improvement | 3.4 | 6.2 | 3.1 | 0.0
  Moderate improvement | 13.6 | 6.2 | 15.6 | 22.2
  Slight improvement | 25.4 | 18.5 | 9.4 | 22.2
  No change | 35.6 | 46.2 | 53.1 | 44.4
  Slight worsening | 18.6 | 16.9 | 12.5 | 0.0
  Moderate worsening | 3.4 | 4.6 | 6.3 | 11.1
  Marked worsening | 0.0 | 1.5 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

28. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 6
Description: Disease evolution compared to the last visit was evaluated by the investigator applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening not done. The GES is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit).
Time Frame: Visit 6 (Month 12)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 54 | 61 | 28 | 9
percentage of participants
  Marked improvement | 5.6 | 1.6 | 10.7 | 11.1
  Moderate improvement | 16.7 | 13.1 | 14.3 | 11.1
  Slight improvement | 22.2 | 19.7 | 17.9 | 22.2
  No change | 29.6 | 41.0 | 39.3 | 55.6
  Slight worsening | 20.4 | 18.0 | 14.3 | 0.0
  Moderate worsening | 3.7 | 6.6 | 3.6 | 0.0
  Marked worsening | 1.9 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

29. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 7
Description: as for outcome 22
Time Frame: Visit 7 (Month 15)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 47 | 52 | 28 | 8
percentage of participants
  Marked improvement | 12.8 | 9.6 | 3.6 | 0.0
  Moderate improvement | 4.3 | 13.5 | 7.1 | 0.0
  Slight improvement | 23.4 | 11.5 | 14.3 | 37.5
  No change | 42.6 | 40.4 | 39.3 | 37.5
  Slight worsening | 12.8 | 21.2 | 25.0 | 12.5
  Moderate worsening | 2.1 | 1.9 | 10.7 | 12.5
  Marked worsening | 2.1 | 1.9 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

30. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 8
Description: as for outcome 22
Time Frame: Visit 8 (Month 18)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 40 | 51 | 28 | 6
percentage of participants
  Marked improvement | 10.0 | 3.9 | 3.6 | 16.7
  Moderate improvement | 5.0 | 11.8 | 17.9 | 0.0
  Slight improvement | 20.0 | 23.5 | 14.3 | 16.7
  No change | 37.5 | 39.2 | 42.9 | 66.7
  Slight worsening | 25.0 | 17.6 | 14.3 | 0.0
  Moderate worsening | 2.5 | 3.9 | 7.1 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

31. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 9
Description: as for outcome 22
Time Frame: Visit 9 (Month 21)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 39 | 49 | 27 | 5
percentage of participants
  Marked improvement | 5.1 | 8.2 | 14.8 | 0.0
  Moderate improvement | 7.7 | 14.3 | 11.1 | 0.0
  Slight improvement | 12.8 | 22.4 | 22.2 | 0.0
  No change | 48.7 | 34.7 | 33.3 | 80.0
  Slight worsening | 23.1 | 18.4 | 7.4 | 20.0
  Moderate worsening | 2.6 | 0.0 | 7.4 | 0.0
  Marked worsening | 0.0 | 2.0 | 3.7 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

32. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 10
Description: as for outcome 28
Time Frame: Visit 10 (Month 24)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 35 | 47 | 25 | 6
percentage of participants
  Marked improvement | 5.7 | 6.4 | 4.0 | 0.0
  Moderate improvement | 8.6 | 12.8 | 8.0 | 0.0
  Slight improvement | 22.9 | 17.0 | 20.0 | 0.0
  No change | 45.7 | 51.1 | 48.0 | 66.7
  Slight worsening | 11.4 | 12.8 | 20.0 | 16.7
  Moderate worsening | 5.7 | 0.0 | 0.0 | 16.7
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

33. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 11
Description: as for outcome 22
Time Frame: Visit 11 (Month 27)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 32 | 44 | 22 | 5
percentage of participants
  Marked improvement | 9.4 | 2.3 | 4.5 | 0.0
  Moderate improvement | 9.4 | 6.8 | 22.7 | 20.0
  Slight improvement | 21.9 | 20.5 | 13.6 | 20.0
  No change | 50.0 | 45.5 | 54.5 | 60.0
  Slight worsening | 6.3 | 15.9 | 4.5 | 0.0
  Moderate worsening | 0.0 | 4.5 | 0.0 | 0.0
  Marked worsening | 0.0 | 2.3 | 0.0 | 0.0
  Not done | 3.1 | 2.3 | 0.0 | 0.0

34. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 12
Description: as for outcome 22
Time Frame: Visit 12 (Month 30)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 30 | 39 | 18 | 4
percentage of participants
  Marked improvement | 6.7 | 5.1 | 0.0 | 0.0
  Moderate improvement | 6.7 | 15.4 | 5.6 | 0.0
  Slight improvement | 33.3 | 25.6 | 11.1 | 25.0
  No change | 33.3 | 43.6 | 61.1 | 75.0
  Slight worsening | 16.7 | 7.7 | 11.1 | 0.0
  Moderate worsening | 0.0 | 2.6 | 11.1 | 0.0
  Marked worsening | 3.3 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

35. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 13
Description: as for outcome 22
Time Frame: Visit 13 (Month 33)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 26 | 30 | 9 | 4
percentage of participants
  Marked improvement | 3.8 | 3.3 | 0.0 | 0.0
  Moderate improvement | 7.7 | 6.7 | 11.1 | 0.0
  Slight improvement | 34.6 | 23.3 | 22.2 | 50.0
  No change | 38.5 | 46.7 | 55.6 | 50.0
  Slight worsening | 15.4 | 16.7 | 11.1 | 0.0
  Moderate worsening | 0.0 | 3.3 | 0.0 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

36. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 14
Description: as for outcome 22
Time Frame: Visit 14 (Month 36)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 15 | 24 | 9 | 0
percentage of participants
  Marked improvement | 13.3 | 4.2 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 0.0 |
  Slight improvement | 33.3 | 16.7 | 11.1 |
  No change | 40.0 | 45.8 | 66.7 |
  Slight worsening | 13.3 | 25.0 | 11.1 |
  Moderate worsening | 0.0 | 8.3 | 11.1 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

37. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 15
Description: as for outcome 22
Time Frame: Visit 15 (Month 39)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 15 | 21 | 7 | 0
percentage of participants
  Marked improvement | 6.7 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 14.3 |
  Slight improvement | 26.7 | 28.6 | 14.3 |
  No change | 46.7 | 61.9 | 57.1 |
  Slight worsening | 6.7 | 9.5 | 14.3 |
  Moderate worsening | 13.3 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

38. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 16
Description: as for outcome 22
Time Frame: Visit 16 (Month 42)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 14 | 18 | 7 | 0
percentage of participants
  Marked improvement | 0.0 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 5.6 | 0.0 |
  Slight improvement | 35.7 | 11.1 | 14.3 |
  No change | 42.9 | 61.1 | 85.7 |
  Slight worsening | 14.3 | 16.7 | 0.0 |
  Moderate worsening | 7.1 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 5.6 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

39. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 17
Description: as for outcome 22
Time Frame: Visit 17 (Month 45)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 13 | 17 | 6 | 0
percentage of participants
  Marked improvement | 7.7 | 11.8 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 16.7 |
  Slight improvement | 38.5 | 17.6 | 0.0 |
  No change | 53.8 | 47.1 | 83.3 |
  Slight worsening | 0.0 | 23.5 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

40. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 18
Description: as for outcome 22
Time Frame: Visit 18 (Month 48)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 13 | 13 | 6 | 0
percentage of participants
  Marked improvement | 7.7 | 15.4 | 16.7 |
  Moderate improvement | 0.0 | 0.0 | 0.0 |
  Slight improvement | 15.4 | 30.8 | 16.7 |
  No change | 46.2 | 38.5 | 50.0 |
  Slight worsening | 30.8 | 15.4 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 16.7 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

41. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 19
Description: as for outcome 22
Time Frame: Visit 19 (Month 51)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 11 | 13 | 5 | 0
percentage of participants
  Marked improvement | 9.1 | 7.7 | 0.0 |
  Moderate improvement | 0.0 | 7.7 | 0.0 |
  Slight improvement | 18.2 | 15.4 | 40.0 |
  No change | 54.5 | 46.2 | 60.0 |
  Slight worsening | 18.2 | 23.1 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

42. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 20
Description: as for outcome 22
Time Frame: Visit 20 (Month 54)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 11 | 12 | 5 | 0
percentage of participants
  Marked improvement | 0.0 | 8.3 | 0.0 |
  Moderate improvement | 9.1 | 0.0 | 0.0 |
  Slight improvement | 18.2 | 16.7 | 0.0 |
  No change | 63.6 | 58.3 | 100.0 |
  Slight worsening | 9.1 | 8.3 | 0.0 |
  Moderate worsening | 0.0 | 8.3 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

43. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 21
Description: as for outcome 22
Time Frame: Visit 21 (Month 57)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 9 | 8 | 5 | 0
percentage of participants
  Marked improvement | 22.2 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 12.5 | 0.0 |
  Slight improvement | 22.2 | 12.5 | 20.0 |
  No change | 55.6 | 62.5 | 80.0 |
  Slight worsening | 0.0 | 12.5 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

44. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 22
Description: as for outcome 22
Time Frame: Visit 22 (Month 60)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 3 | 4 | 5 | 0
percentage of participants
  Marked improvement | 33.3 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 20.0 |
  Slight improvement | 0.0 | 0.0 | 20.0 |
  No change | 33.3 | 75.0 | 60.0 |
  Slight worsening | 33.3 | 0.0 | 0.0 |
  Moderate worsening | 0.0 | 25.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

45. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 23
Description: as for outcome 22
Time Frame: Visit 23 (Month 63)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 2 | 1 | 5 | 0
percentage of participants
  Marked improvement | 0.0 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 20.0 |
  Slight improvement | 50.0 | 100.0 | 20.0 |
  No change | 50.0 | 0.0 | 40.0 |
  Slight worsening | 0.0 | 0.0 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 20.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

46. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 24
Description: as for outcome 22
Time Frame: Visit 24 (Month 66)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 1 | 0 | 5 | 0
percentage of participants
  Marked improvement | 0.0 |  | 20.0 |
  Moderate improvement | 0.0 |  | 0.0 |
  Slight improvement | 0.0 |  | 0.0 |
  No change | 100.0 |  | 80.0 |
  Slight worsening | 0.0 |  | 0.0 |
  Moderate worsening | 0.0 |  | 0.0 |
  Marked worsening | 0.0 |  | 0.0 |
  Not done | 0.0 |  | 0.0 |

47. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 25
Description: as for outcome 22
Time Frame: Visit 25 (Month 69)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

48. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 26
Description: as for outcome 22
Time Frame: Visit 26 (Month 72)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 25.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

49. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 27
Description: as for outcome 22
Time Frame: Visit 27 (Month 75)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 25.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

50. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 28
Description: as for outcome 22
Time Frame: Visit 28 (Month 78)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

51. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 29
Description: as for outcome 22
Time Frame: Visit 29 (Month 81)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 25.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

52. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 30
Description: as for outcome 22
Time Frame: Visit 30 (Month 84)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

53. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 31
Description: as for outcome 22
Time Frame: Visit 31 (Month 87)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 2 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

54. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Withdrawal Visit
Description: as for outcome 22
Time Frame: Withdrawal visit (up to Month 90)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 17 | 14 | 5 | 4
percentage of participants
  Marked improvement | 5.9 | 0.0 | 0.0 | 0.0
  Moderate improvement | 5.9 | 7.1 | 0.0 | 0.0
  Slight improvement | 5.9 | 0.0 | 20.0 | 25.0
  No change | 41.2 | 50.0 | 0.0 | 75.0
  Slight worsening | 11.8 | 35.7 | 60.0 | 0.0
  Moderate worsening | 23.5 | 0.0 | 20.0 | 0.0
  Marked worsening | 5.9 | 7.1 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

55. Secondary Outcome: Percentage of Subjects in Categories of Investigator's Rating of Change to Previous Visit in Global Evaluation Scale at Final Visit
Description: as for outcome 22
Time Frame: Final visit (up to Month 90)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 69 | 81 | 41 | 13
percentage of participants
  Marked improvement | 4.3 | 3.7 | 2.4 | 7.7
  Moderate improvement | 11.6 | 6.2 | 17.1 | 0.0
  Slight improvement | 23.2 | 9.9 | 14.6 | 7.7
  No change | 36.2 | 61.7 | 51.2 | 69.2
  Slight worsening | 17.4 | 9.9 | 4.9 | 15.4
  Moderate worsening | 4.3 | 6.2 | 9.8 | 0.0
  Marked worsening | 1.4 | 0.0 | 0.0 | 0.0
  Not done | 1.4 | 2.5 | 0.0 | 0.0

56. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 1
Description: Disease evolution compared to the last visit was evaluated by the parent/legal guardian applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening, not done. The GES is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit). The reference time point for Visit 1 is in the respective feeder study of the participant.
Time Frame: Visit 1 (Screening Visit (Week 0))
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 78 | 89 | 41 | 14
percentage of participants
  Marked improvement | 12.8 | 18.0 | 29.3 | 0.0
  Moderate improvement | 16.7 | 15.7 | 14.6 | 0.0
  Slight improvement | 17.9 | 19.1 | 14.6 | 0.0
  No change | 41.0 | 38.2 | 24.4 | 92.9
  Slight worsening | 7.7 | 7.9 | 17.1 | 7.1
  Moderate worsening | 3.8 | 0.0 | 0.0 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 1.1 | 0.0 | 0.0

57. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 1
Description: Disease evolution compared to the last visit was evaluated by the parent/legal guardian applying following categories: Marked improvement, moderate improvement, slight improvement, no change, slight worsening, moderate worsening, marked worsening, not done. The GES is a 7-point scale wherein 7 categories are ranked from 1 (marked improvement from previous visit) to 7 (marked worsening from previous visit).
Time Frame: Titration Visit 1 (Week 2)
Population: as for outcome 21
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 74 | 82 | 0 | 0
percentage of participants
  Marked improvement | 17.6 | 11.0 |  |
  Moderate improvement | 18.9 | 11.0 |  |
  Slight improvement | 32.4 | 17.1 |  |
  No change | 25.7 | 48.8 |  |
  Slight worsening | 4.1 | 8.5 |  |
  Moderate worsening | 0.0 | 1.2 |  |
  Marked worsening | 0.0 | 0.0 |  |
  Not done | 1.4 | 2.4 |  |

58. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 2
Description: as for outcome 57
Time Frame: Titration Visit 2 (Week 4)
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 75 | 84 | 0 | 0
percentage of participants
  Marked improvement | 17.3 | 16.7 |  |
  Moderate improvement | 16.0 | 10.7 |  |
  Slight improvement | 20.0 | 15.5 |  |
  No change | 36.0 | 39.3 |  |
  Slight worsening | 6.7 | 15.5 |  |
  Moderate worsening | 2.7 | 1.2 |  |
  Marked worsening | 0.0 | 0.0 |  |
  Not done | 1.3 | 1.2 |  |

59. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Titration Visit 3
Description: as for outcome 57
Time Frame: Titration Visit 3 (Week 6)
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 67 | 73 | 0 | 0
percentage of participants
  Marked improvement | 10.4 | 4.1 |  |
  Moderate improvement | 9.0 | 12.3 |  |
  Slight improvement | 20.9 | 27.4 |  |
  No change | 43.3 | 41.1 |  |
  Slight worsening | 9.0 | 8.2 |  |
  Moderate worsening | 3.0 | 4.1 |  |
  Marked worsening | 1.5 | 1.4 |  |
  Not done | 3.0 | 1.4 |  |

60. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 2
Description: as for outcome 57
Time Frame: Visit 2 (Month 2)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 73 | 84 | 39 | 12
percentage of participants
  Marked improvement | 6.8 | 13.1 | 25.6 | 16.7
  Moderate improvement | 17.8 | 11.9 | 15.4 | 8.3
  Slight improvement | 21.9 | 16.7 | 20.5 | 41.7
  No change | 30.1 | 45.2 | 17.9 | 8.3
  Slight worsening | 17.8 | 4.8 | 17.9 | 0.0
  Moderate worsening | 2.7 | 4.8 | 2.6 | 8.3
  Marked worsening | 2.7 | 1.2 | 0.0 | 16.7
  Not done | 0.0 | 2.4 | 0.0 | 0.0

61. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 3
Description: as for outcome 57
Time Frame: Visit 3 (Month 4)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 68 | 77 | 38 | 10
percentage of participants
  Marked improvement | 8.8 | 6.5 | 18.4 | 20.0
  Moderate improvement | 5.9 | 6.5 | 15.8 | 20.0
  Slight improvement | 16.2 | 13.0 | 18.4 | 20.0
  No change | 38.2 | 48.1 | 36.8 | 30.0
  Slight worsening | 19.1 | 22.1 | 7.9 | 10.0
  Moderate worsening | 10.3 | 3.9 | 2.6 | 0.0
  Marked worsening | 1.5 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

62. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 4
Description: as for outcome 57
Time Frame: Visit 4 (Month 6)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 63 | 75 | 35 | 10
percentage of participants
  Marked improvement | 4.8 | 8.0 | 20.0 | 20.0
  Moderate improvement | 7.9 | 6.7 | 14.3 | 0.0
  Slight improvement | 22.2 | 29.3 | 5.7 | 20.0
  No change | 39.7 | 33.3 | 37.1 | 50.0
  Slight worsening | 19.0 | 17.3 | 17.1 | 10.0
  Moderate worsening | 4.8 | 5.3 | 5.7 | 0.0
  Marked worsening | 1.6 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

63. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 5
Description: as for outcome 57
Time Frame: Visit 5 (Month 9)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 59 | 65 | 32 | 9
percentage of participants
  Marked improvement | 6.8 | 10.8 | 9.4 | 11.1
  Moderate improvement | 10.2 | 6.2 | 9.4 | 33.3
  Slight improvement | 25.4 | 12.3 | 9.4 | 11.1
  No change | 33.9 | 46.2 | 50.0 | 33.3
  Slight worsening | 20.3 | 15.4 | 9.4 | 0.0
  Moderate worsening | 0.0 | 6.2 | 12.5 | 11.1
  Marked worsening | 3.4 | 3.1 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

64. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 6
Description: as for outcome 57
Time Frame: Visit 6 (Month 12)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 54 | 61 | 28 | 9
percentage of participants
  Marked improvement | 7.4 | 8.2 | 14.3 | 11.1
  Moderate improvement | 9.3 | 13.1 | 14.3 | 11.1
  Slight improvement | 25.9 | 23.0 | 14.3 | 22.2
  No change | 33.3 | 34.4 | 39.3 | 55.6
  Slight worsening | 18.5 | 11.5 | 14.3 | 0.0
  Moderate worsening | 3.7 | 8.2 | 3.6 | 0.0
  Marked worsening | 1.9 | 1.6 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

65. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 7
Description: as for outcome 57
Time Frame: Visit 7 (Month 15)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 47 | 52 | 28 | 8
percentage of participants
  Marked improvement | 10.6 | 19.2 | 7.1 | 0.0
  Moderate improvement | 10.6 | 9.6 | 7.1 | 0.0
  Slight improvement | 23.4 | 7.7 | 10.7 | 37.5
  No change | 29.8 | 40.4 | 42.9 | 37.5
  Slight worsening | 19.1 | 15.4 | 25.0 | 12.5
  Moderate worsening | 4.3 | 3.8 | 3.6 | 0.0
  Marked worsening | 2.1 | 1.9 | 3.6 | 12.5
  Not done | 0.0 | 1.9 | 0.0 | 0.0

66. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 8
Description: as for outcome 57
Time Frame: Visit 8 (Month 18)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 40 | 51 | 28 | 6
percentage of participants
  Marked improvement | 5.0 | 15.7 | 7.1 | 16.7
  Moderate improvement | 7.5 | 9.8 | 14.3 | 0.0
  Slight improvement | 17.5 | 17.6 | 14.3 | 16.7
  No change | 45.0 | 35.3 | 42.9 | 66.7
  Slight worsening | 22.5 | 15.7 | 10.7 | 0.0
  Moderate worsening | 2.5 | 3.9 | 10.7 | 0.0
  Marked worsening | 0.0 | 2.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

67. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 9
Description: as for outcome 57
Time Frame: Visit 9 (Month 21)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 39 | 49 | 27 | 5
percentage of participants
  Marked improvement | 10.3 | 12.2 | 18.5 | 0.0
  Moderate improvement | 7.7 | 10.2 | 7.4 | 0.0
  Slight improvement | 10.3 | 14.3 | 22.2 | 40.0
  No change | 56.4 | 53.1 | 33.3 | 40.0
  Slight worsening | 10.3 | 6.1 | 3.7 | 0.0
  Moderate worsening | 5.1 | 2.0 | 11.1 | 20.0
  Marked worsening | 0.0 | 2.0 | 3.7 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

68. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 10
Description: as for outcome 57
Time Frame: Visit 10 (Month 24)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 35 | 47 | 25 | 6
percentage of participants
  Marked improvement | 8.6 | 8.5 | 12.0 | 0.0
  Moderate improvement | 5.7 | 8.5 | 4.0 | 0.0
  Slight improvement | 22.9 | 21.3 | 20.0 | 16.7
  No change | 42.9 | 48.9 | 40.0 | 66.7
  Slight worsening | 11.4 | 10.6 | 20.0 | 0.0
  Moderate worsening | 5.7 | 2.1 | 0.0 | 16.7
  Marked worsening | 2.9 | 0.0 | 4.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

69. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 11
Description: as for outcome 57
Time Frame: Visit 11 (Month 27)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 32 | 44 | 22 | 5
percentage of participants
  Marked improvement | 9.4 | 9.1 | 9.1 | 0.0
  Moderate improvement | 9.4 | 4.5 | 22.7 | 20.0
  Slight improvement | 18.8 | 18.2 | 9.1 | 20.0
  No change | 53.1 | 45.5 | 54.5 | 40.0
  Slight worsening | 6.3 | 11.4 | 4.5 | 20.0
  Moderate worsening | 0.0 | 6.8 | 0.0 | 0.0
  Marked worsening | 0.0 | 2.3 | 0.0 | 0.0
  Not done | 3.1 | 2.3 | 0.0 | 0.0

70. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 12
Description: as for outcome 57
Time Frame: Visit 12 (Month 30)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 30 | 39 | 18 | 4
percentage of participants
  Marked improvement | 6.7 | 7.7 | 0.0 | 0.0
  Moderate improvement | 13.3 | 12.8 | 11.1 | 0.0
  Slight improvement | 26.7 | 20.5 | 5.6 | 25.0
  No change | 33.3 | 48.7 | 55.6 | 75.0
  Slight worsening | 16.7 | 5.1 | 16.7 | 0.0
  Moderate worsening | 3.3 | 2.6 | 11.1 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 2.6 | 0.0 | 0.0

71. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 13
Description: as for outcome 57
Time Frame: Visit 13 (Month 33)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 26 | 30 | 9 | 4
percentage of participants
  Marked improvement | 7.7 | 3.3 | 0.0 | 0.0
  Moderate improvement | 23.1 | 6.7 | 11.1 | 0.0
  Slight improvement | 15.4 | 23.3 | 22.2 | 25.0
  No change | 38.5 | 46.7 | 55.6 | 75.0
  Slight worsening | 15.4 | 16.7 | 11.1 | 0.0
  Moderate worsening | 0.0 | 3.3 | 0.0 | 0.0
  Marked worsening | 0.0 | 0.0 | 0.0 | 0.0
  Not done | 0.0 | 0.0 | 0.0 | 0.0

72. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 14
Description: as for outcome 57
Time Frame: Visit 14 (Month 36)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 15 | 24 | 9 | 0
percentage of participants
  Marked improvement | 20.0 | 4.2 | 0.0 |
  Moderate improvement | 0.0 | 4.2 | 0.0 |
  Slight improvement | 26.7 | 12.5 | 11.1 |
  No change | 40.0 | 50.0 | 66.7 |
  Slight worsening | 13.3 | 20.8 | 22.2 |
  Moderate worsening | 0.0 | 4.2 | 0.0 |
  Marked worsening | 0.0 | 4.2 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

73. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 15
Description: as for outcome 57
Time Frame: Visit 15 (Month 39)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 15 | 21 | 7 | 0
percentage of participants
  Marked improvement | 6.7 | 0.0 | 0.0 |
  Moderate improvement | 6.7 | 0.0 | 14.3 |
  Slight improvement | 40.0 | 28.6 | 14.3 |
  No change | 40.0 | 52.4 | 57.1 |
  Slight worsening | 6.7 | 9.5 | 14.3 |
  Moderate worsening | 0.0 | 4.8 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 4.8 | 0.0 |

74. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 16
Description: as for outcome 57
Time Frame: Visit 16 (Month 42)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 14 | 18 | 7 | 0
percentage of participants
  Marked improvement | 7.1 | 0.0 | 0.0 |
  Moderate improvement | 21.4 | 0.0 | 0.0 |
  Slight improvement | 14.3 | 16.7 | 28.6 |
  No change | 35.7 | 55.6 | 71.4 |
  Slight worsening | 14.3 | 22.2 | 0.0 |
  Moderate worsening | 7.1 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 5.6 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

75. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 17
Description: as for outcome 57
Time Frame: Visit 17 (Month 45)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 13 | 17 | 6 | 0
percentage of participants
  Marked improvement | 15.4 | 11.8 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 16.7 |
  Slight improvement | 38.5 | 23.5 | 0.0 |
  No change | 46.2 | 41.2 | 83.3 |
  Slight worsening | 0.0 | 17.6 | 0.0 |
  Moderate worsening | 0.0 | 5.9 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

76. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 18
Description: as for outcome 57
Time Frame: Visit 18 (Month 48)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 13 | 13 | 6 | 0
percentage of participants
  Marked improvement | 0.0 | 15.4 | 16.7 |
  Moderate improvement | 0.0 | 7.7 | 0.0 |
  Slight improvement | 23.1 | 23.1 | 16.7 |
  No change | 38.5 | 38.5 | 50.0 |
  Slight worsening | 38.5 | 15.4 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 16.7 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

77. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 19
Description: as for outcome 57
Time Frame: Visit 19 (Month 51)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 11 | 13 | 5 | 0
percentage of participants
  Marked improvement | 9.1 | 7.7 | 0.0 |
  Moderate improvement | 0.0 | 7.7 | 0.0 |
  Slight improvement | 27.3 | 23.1 | 40.0 |
  No change | 45.5 | 38.5 | 60.0 |
  Slight worsening | 18.2 | 23.1 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

78. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 20
Description: as for outcome 57
Time Frame: Visit 20 (Month 54)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 11 | 12 | 5 | 0
percentage of participants
  Marked improvement | 9.1 | 8.3 | 0.0 |
  Moderate improvement | 9.1 | 0.0 | 0.0 |
  Slight improvement | 9.1 | 16.7 | 0.0 |
  No change | 63.6 | 66.7 | 100.0 |
  Slight worsening | 9.1 | 0.0 | 0.0 |
  Moderate worsening | 0.0 | 8.3 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

79. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 21
Description: as for outcome 57
Time Frame: Visit 21 (Month 57)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 9 | 8 | 5 | 0
percentage of participants
  Marked improvement | 22.2 | 0.0 | 0.0 |
  Moderate improvement | 0.0 | 0.0 | 20.0 |
  Slight improvement | 22.2 | 37.5 | 20.0 |
  No change | 55.6 | 50.0 | 60.0 |
  Slight worsening | 0.0 | 12.5 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

80. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 22
Description: as for outcome 57
Time Frame: Visit 22 (Month 60)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 3 | 4 | 5 | 0
percentage of participants
  Marked improvement | 33.3 | 0.0 | 20.0 |
  Moderate improvement | 0.0 | 0.0 | 0.0 |
  Slight improvement | 0.0 | 0.0 | 20.0 |
  No change | 33.3 | 75.0 | 60.0 |
  Slight worsening | 33.3 | 0.0 | 0.0 |
  Moderate worsening | 0.0 | 25.0 | 0.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

81. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 23
Description: as for outcome 57
Time Frame: Visit 23 (Month 63)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 2 | 1 | 5 | 0
percentage of participants
  Marked improvement | 0.0 | 0.0 | 0.0 |
  Moderate improvement | 50.0 | 0.0 | 20.0 |
  Slight improvement | 0.0 | 100.0 | 20.0 |
  No change | 50.0 | 0.0 | 40.0 |
  Slight worsening | 0.0 | 0.0 | 0.0 |
  Moderate worsening | 0.0 | 0.0 | 20.0 |
  Marked worsening | 0.0 | 0.0 | 0.0 |
  Not done | 0.0 | 0.0 | 0.0 |

82. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 24
Description: as for outcome 57
Time Frame: Visit 24 (Month 66)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 1 | 0 | 5 | 0
percentage of participants
  Marked improvement | 0.0 |  | 20.0 |
  Moderate improvement | 0.0 |  | 0.0 |
  Slight improvement | 0.0 |  | 0.0 |
  No change | 100.0 |  | 80.0 |
  Slight worsening | 0.0 |  | 0.0 |
  Moderate worsening | 0.0 |  | 0.0 |
  Marked worsening | 0.0 |  | 0.0 |
  Not done | 0.0 |  | 0.0 |

83. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 25
Description: as for outcome 57
Time Frame: Visit 25 (Month 69)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

84. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 26
Description: as for outcome 57
Time Frame: Visit 26 (Month 72)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 25.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

85. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 27
Description: as for outcome 57
Time Frame: Visit 27 (Month 75)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 25.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

86. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 28
Description: as for outcome 57
Time Frame: Visit 28 (Month 78)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

87. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 29
Description: as for outcome 57
Time Frame: Visit 29 (Month 81)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 75.0 |
  Slight worsening |  |  | 25.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

88. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 30
Description: as for outcome 57
Time Frame: Visit 30 (Month 84)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 4 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

89. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Visit 31
Description: as for outcome 57
Time Frame: Visit 31 (Month 87)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 0 | 0 | 2 | 0
percentage of participants
  Marked improvement |  |  | 0.0 |
  Moderate improvement |  |  | 0.0 |
  Slight improvement |  |  | 0.0 |
  No change |  |  | 100.0 |
  Slight worsening |  |  | 0.0 |
  Moderate worsening |  |  | 0.0 |
  Marked worsening |  |  | 0.0 |
  Not done |  |  | 0.0 |

90. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Withdrawal Visit
Description: as for outcome 57
Time Frame: Withdrawal visit (up to Month 90)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 17 | 14 | 5 | 4
percentage of participants
  Marked improvement | 5.9 | 7.1 | 0.0 | 0.0
  Moderate improvement | 0.0 | 0.0 | 0.0 | 0.0
  Slight improvement | 5.9 | 0.0 | 20.0 | 25.0
  No change | 41.2 | 42.9 | 40.0 | 75.0
  Slight worsening | 29.4 | 21.4 | 20.0 | 0.0
  Moderate worsening | 17.6 | 14.3 | 20.0 | 0.0
  Marked worsening | 0.0 | 7.1 | 0.0 | 0.0
  Not done | 0.0 | 7.1 | 0.0 | 0.0

91. Secondary Outcome: Percentage of Subjects in Categories of Parent/Legal Guardian's Rating of Change to Previous Visit in Global Evaluation Scale at Final Visit
Description: as for outcome 57
Time Frame: Final visit (up to Month 90)
Population: Only subjects with available data for disease evolution compared to the previous visit are included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
Number analyzed (Participants) | 69 | 81 | 41 | 13
percentage of participants
  Marked improvement | 8.7 | 7.4 | 4.9 | 7.7
  Moderate improvement | 14.5 | 8.6 | 12.2 | 0.0
  Slight improvement | 15.9 | 6.2 | 14.6 | 7.7
  No change | 34.8 | 58.0 | 51.2 | 69.2
  Slight worsening | 17.4 | 13.6 | 4.9 | 15.4
  Moderate worsening | 0.0 | 3.7 | 4.9 | 0.0
  Marked worsening | 5.8 | 1.2 | 7.3 | 0.0
  Not done | 2.9 | 1.2 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose in N157 to End of the Study (up to 7.5 years)
Description: Adverse Events refer to the Safety Population, including all randomized subjects who received at least one dose of study medication.
Arm/Group | N159 PBO/LEV | N159 LEV/LEV | N01010+N151 LEV/LEV | N01052 LEV/LEV
All-Cause Mortality (participants affected / at risk) | 0/79 | 1/89 | 0/41 | 0/14
Serious Adverse Events (participants affected / at risk) | 20/79 | 35/89 | 12/41 | 7/14
Other Adverse Events (participants affected / at risk) | 77/79 | 86/89 | 41/41 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N159 PBO/LEV (N=79) | N159 LEV/LEV (N=89) | N01010+N151 LEV/LEV (N=41) | N01052 LEV/LEV (N=14)
Asthenia (General disorders) | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 1 | 1 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Infection (General disorders) | 0 | 0 | 0 | 1
Infection bacterial (General disorders) | 0 | 0 | 1 | 0
Overdose (General disorders) | 1 | 1 | 0 | 0
Reaction unevaluable (General disorders) | 0 | 1 | 0 | 0
Heart arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Hemorrhage (Cardiac disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fecal impaction (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gasteroenteritis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Increased salivation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach atony (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Endocrine disorders) | 0 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Albuminuria (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Musculoskeletal congenital anomaly (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myasthenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Antisocial reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Nervous system disorders) | 0 | 1 | 0 | 0
Apathy (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 9 | 7 | 2 | 4
Depression (Nervous system disorders) | 1 | 2 | 0 | 0
Intracranial hypertension (Nervous system disorders) | 0 | 0 | 1 | 0
Nervousness (Nervous system disorders) | 0 | 1 | 0 | 0
Personality disorder (Nervous system disorders) | 0 | 3 | 0 | 0
Psychosis (Nervous system disorders) | 1 | 1 | 0 | 0
Pschychotic depression (Nervous system disorders) | 1 | 0 | 0 | 0
Schizophrenic reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 1 | 0 | 1
Status epilepticus partial (Nervous system disorders) | 1 | 0 | 1 | 0
Procedure diagnostic epilepsy (Investigations) | 2 | 9 | 1 | 0
Procedure diagnostic (Investigations) | 1 | 1 | 2 | 0
Procedure therapeutic epilepsy (Investigations) | 2 | 8 | 5 | 0
Procedure therapeutic (Investigations) | 1 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Kidney calculus (Renal and urinary disorders) | 0 | 0 | 1 | 1
Pyelonephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urogenital disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N159 PBO/LEV (N=79) | N159 LEV/LEV (N=89) | N01010+N151 LEV/LEV (N=41) | N01052 LEV/LEV (N=14)
Abdominal pain (General disorders) | 9 | 11 | 7 | 1
Accidental injury (General disorders) | 18 | 26 | 9 | 3
Allergic reaction (General disorders) | 8 | 8 | 4 | 1
Asthenia (General disorders) | 10 | 7 | 4 | 0
Drug level increased (General disorders) | 0 | 1 | 1 | 1
Fever (General disorders) | 24 | 23 | 9 | 7
Flu syndrome (General disorders) | 8 | 9 | 5 | 0
Headache (General disorders) | 19 | 23 | 15 | 0
Hostility (General disorders) | 7 | 12 | 6 | 0
Infection (General disorders) | 46 | 48 | 20 | 10
Infection fungal (General disorders) | 0 | 1 | 2 | 1
Pain (General disorders) | 6 | 16 | 7 | 1
Sepsis (General disorders) | 1 | 0 | 0 | 1
Viral infection (General disorders) | 8 | 5 | 6 | 1
Electrocardiogram abnormal (Cardiac disorders) | 0 | 1 | 3 | 0
Anorexia (Gastrointestinal disorders) | 7 | 8 | 6 | 4
Constipation (Gastrointestinal disorders) | 8 | 6 | 4 | 2
Diarrhea (Gastrointestinal disorders) | 6 | 12 | 9 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 3 | 0
Gamma glutamyl transpeptidase increased (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 14 | 8 | 4 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Hemorrhagic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Increased salivation (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 5 | 3 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 15 | 16 | 11 | 4
Accerlerated sexual maturity (Endocrine disorders) | 1 | 0 | 0 | 1
Ecchymosis (Blood and lymphatic system disorders) | 3 | 5 | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 6 | 1
Creatine phosphokinase increased (Metabolism and nutrition disorders) | 2 | 6 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Sgot increased (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 6 | 7 | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 5 | 4 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Myasthenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 1
Strabismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Agitation (Nervous system disorders) | 5 | 4 | 3 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 4 | 0
Anxiety (Nervous system disorders) | 2 | 4 | 3 | 0
Ataxia (Nervous system disorders) | 1 | 2 | 1 | 1
CNS congenital anomaly (Nervous system disorders) | 0 | 0 | 0 | 1
Confusion (Nervous system disorders) | 1 | 3 | 3 | 0
Convulsion (Nervous system disorders) | 8 | 12 | 2 | 2
Depression (Nervous system disorders) | 3 | 5 | 2 | 0
Dizziness (Nervous system disorders) | 4 | 11 | 3 | 0
Emotional lability (Nervous system disorders) | 9 | 4 | 4 | 0
Hyperkinesia (Nervous system disorders) | 2 | 7 | 3 | 1
Insomnia (Nervous system disorders) | 11 | 14 | 6 | 0
Nervousness (Nervous system disorders) | 1 | 5 | 14 | 2
Paresthesia (Nervous system disorders) | 3 | 0 | 4 | 0
Personality disorder (Nervous system disorders) | 11 | 12 | 5 | 0
Psychosis (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 20 | 18 | 10 | 3
Speech disorder (Nervous system disorders) | 3 | 2 | 1 | 2
Thinking abnormal (Nervous system disorders) | 6 | 10 | 2 | 0
Procedure therapeutic (Investigations) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2
Cough increased (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 1 | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 | 20 | 11 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 10 | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 5 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 6 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Contact dermatitis (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 9 | 7 | 4
Conjunctivitis (Eye disorders) | 4 | 3 | 2 | 2
Ear disorder (Ear and labyrinth disorders) | 1 | 5 | 1 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 5 | 3 | 0
Otitis media (Ear and labyrinth disorders) | 17 | 19 | 9 | 7
Urinary tract infection (Renal and urinary disorders) | 2 | 4 | 3 | 0
Urine abnormability (Renal and urinary disorders) | 4 | 4 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days